CLINICAL TRIAL: NCT04363450
Title: Hydroxychloroquine as Primary Prophylaxis for COVID-19 in Healthcare Workers (HCQPreP)
Brief Title: Hydroxychloroquine as Prophylaxis for COVID-19 in Healthcare Workers (HCQPreP)
Acronym: HCQPreP
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Louisiana State University Health Sciences Center in New Orleans (Other)
Collaborators: Lafayette General Health (Other); University of Louisiana at Lafayette (Other)
Responsible Party: Principal Investigator, Ann Chauffe, DO, MPH, Louisiana State University Health Sciences Center in New Orleans
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: LSU NO HSC IRB 20-050
Record Dates: First submitted 2020-04-23; First posted 2020-04-27 (Actual); Last update posted 2020-09-02 (Actual); Status verified 2020-08

CONDITIONS: COVID-19; Corona Virus Infection; Wuhan Coronavirus; Prophylaxis; Healthcare Worker; Sars-CoV2; Hydroxychloroquine
Keywords: COVID-19; COVID-19 Prophylaxis; Healthcare Workers; SARS-COV-2; Hydroxychloroquine
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — Hydroxychloroquine

STUDY DESIGN:
Intervention Model Description: Randomized, placebo-controlled, double-blind study with 1:1 randomization of hydroxychloroquine to placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants will be randomized to the investigational drug (hydroxychloroquine) or placebo. Both will have identical appearance and will be taken at the same dosing interval. The administration of the drug and assessment will be blinded. After final analysis, study arms will be unmasked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Hydroxychloroquine (Experimental): Hydroxychloroquine loading dose will be given as 400mg for two doses 12 hours apart. This will then be followed by maintenance dosing of 200mg twice weekly for the remainder of the trial.
  Interventions: Drug: Hydroxychloroquine
- Placebo (Placebo Comparator): An identical placebo will be administered on an identical dosing interval and frequency.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Hydroxychloroquine — Hydroxychloroquine loading 400mg (2 capsules) twice 12 hours apart followed by 200mg (1 capsule) twice weekly
  Other Names: HCQ PreP
  Arms: Hydroxychloroquine
Drug: Placebo — Loading dose of two placebo capsules twice 12 hours apart followed by 1 capsule twice weekly
  Arms: Placebo

SUMMARY:
This a double-blind, randomized, placebo-controlled clinical trial to determine if primary prophylaxis with hydroxychloroquine in healthcare workers reduces symptomatic COVID-19 infection. Healthcare workers will be randomized at a 1:1 allocation between intervention and placebo arms and followed for 12 weeks. This study will enroll up to 1,700 participates in Lafayette, Louisiana. The primary outcome will number of symptomatic COVID-19 infections. Secondary endpoints included number of days healthcare workers are absent from work and rate of severe infection.

DETAILED DESCRIPTION:
The study is a double blind placebo controlled at two hospitals in Lafayette, Louisiana aiming to enroll 1700 participants with a 1:1 randomization. The HCQ dose in 400mg twice on day 1, then 200mg twice weekly. The primary outcome variable is development of symptomatic COVID-19 infection. The secondary objectives are number of days absent from work due to symptomatic COVID-19 infection and rate of severe disease due to COVID-19 (hypoxia in setting of >50% lung involvement on chest imaging, respiratory failure, shock or end-organ damage). The study will enroll participants for four weeks with and plan to treat with hydroxychloroquine versus placebo for a total of 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Healthcare or Hospital Worker who has direct patient contact
3. Willing to participate in the research.
4. Able to understand and sign the informed consent form

Exclusion Criteria:

1. Age < 18 years
2. History of ventricular arrhythmia or use of Class IA, IC and III anti-arrhythmics
3. Known prolonged QTc interval
4. History of retinal disease
5. Kidney failure with GFR <10%
6. Chronic hepatic disease w/ Child-Pugh class B or C
7. Hypersensitivity to chloroquine or hydroxychloroquine
8. Currently taking chloroquine or hydroxychloroquine
9. Unwilling to participate
10. Unable to understand and/or sign the informed consent form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1700 (Estimated)
Dates: Start 2020-04-27 (Actual); Primary Completion 2021-03-31 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of symptomatic COVID-19 infection in healthcare workers | 12 weeks
  Number of participants who develop symptoms of COVID-19 in the setting of a positive COVID-19 assay

SECONDARY OUTCOMES:
Absenteeism from work due to COVID-19 | 12 weeks
  Number of days healthcare workers are absent from work due to symptomatic COVID-19 infection
Severity of COVID-19 infection | 12 weeks
  Rate of severe COVID-19 infection in healthcare works (hypoxia in setting of chest imaging >50% lung involvement, respiratory failure, end organ damage or shock)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Lafayette General Medical Center, Lafayette, Louisiana
  - University Hospital and Clinics, Lafayette, Louisiana

IPD SHARING:
Plan to Share IPD: No